



sculty of Medicine, University of Indonesia-Central Java Hospital

### **EXPLANATION SHEET TO PROSPECTIVE SUBJECTS**

I, Dr. Melinda Harini, Sp.KFR-K from the Department of Medical Rehabilitation, CIPTO National Hospital MANGUNKUSUMO will conduct research entitled Effectiveness of Adding *Virtual* Training

The Reality of Early Mobilization Program on Quality of Life of Patients in Integrated Geriatric Acute Ward.

I will provide information to (Sir/Madam/Brother) regarding this research and invite you to participate. (Sir/Madam/Brother) to be part of this research.

You can participate in this research by signing this form. If Sir/Madam/Brother agrees to participate in this research, Sir/Madam/Brother can at any time free to withdraw from this research. If you refuse to participate or withdraw from the research this decision will not affect your relationship with me and will not affect you. impact on the services provided at this hospital.

If you do not understand any statement in this form, you can ask me.

### 1. Research objectives

To determine the effectiveness of adding VR training to the activity process carried out during treatment in hospital on the quality of life of patients in integrated elderly inpatient rooms. VR is a technology that allows users to interact with a computer-simulated environment.

# 2. Participation in research

If you decide to participate in this research, you

will act as a limited user target for the VR system that has been developed (already

passing trials that test the ease and effectiveness of a digital product or system that can

used by the user). First, you will be interviewed by a doctor, then

Sir/Madam/Brother, you are requested to use the VR system in carrying out shopping activities and

Follow the instructions given. After completion, you will be given several questionnaires.

to be filled in according to the experience felt when using the VR system. This research took
time approximately 30 minutes.





Faculty of Medicine, University of Indonesia-Central Java Hospita

# 3. Reasons for choosing Mr/Mrs/Sibling

We will take part in this research if you have stated your willingness and sign the consent form, age more than or equal to 60 years, and meet the criteria.

Our research subjects are:

Inclusion Criteria:

- Able to understand instructions and commands Able

  to move upper limbs against gravity (upper limb strength is more than or equal to 3) or at least the patient is able to sit

  beside the bed independently or with assistance
- Can communicate adequately receptively and expressively
- Ha<u>ving various disease conditions that interact to cause complications in medical management more than</u> or equal to 5

Ladies and gentlemen who are willing to participate in the research program will sign a letter of consent.

### **Exclusion Criteria:**

- Complaints of dizziness when the view or focus of vision changes
- Discharge plan from the integrated elderly inpatient ward before 1 week
- Having serious mental and social problems
- · Heavy burden on caregivers

## 4. Research procedures

| to participate in the research after the researcher explains to you the research subjects |
|---|
| regarding the objectives, benefits, and procedures of the research. You will undergo an interview process. |
| and a brief physical examination (blood pressure, heart rate, respiratory rate, blood oxygen levels, |
| assessment of quality of life, level of physical activity intensity using ratio scale measurements, lactate examination |
| blood, measuring the level of independence in basic daily activities, measuring the reduction in |
| the ability and function of adjustment resulting from a decline in the function of the body's systems and |
| measuring the decrease in muscle size and strength) before rehabilitation is given to |
| get your initial grades, sir/madam/brother. |
| Sir/Madam/Brother/Sir, you will be prepared to use the Virtual Reality (VR) device that has been |
| programmed to follow the assessment procedures according to the research protocol. The attending physician |
| responsible for conducting inspections to assess the conditions that are permitted and not permitted during |
| using VR. After receiving an explanation, you will familiarize yourself with the OculusR equipment, which is part of the |
| VR, and adjust the view seen from the VR. |
| Sir/Madam/Brother start the game and complete the VRAGMENT activities step by step. |
| Throughout the game, the caregiver and DPJP may provide playing instructions and feedback to the child. |
| encourage Mr/Mrs/Brother. The duration of play is recorded, the patient's target is to play for 30 minutes continuously |





### **Health Research Ethics Committee**

| | Continuously or according to patient tolerance. Exercises were performed 5 times a week. During the study |
|---|---|
| | Using VR, you will be accompanied by trained personnel for your safety. |
| | Once completed, you will be assessed again (blood pressure, heart rate, breathing rate and levels |
| | oxygen in the blood). |
| | Ladies and Gentlemen who participate in the research will be re-examined for assessment (quality of life, level of |
| | intensity of physical activity using ratio scale measurements, blood lactate examination, measuring the level of |
| | independence in basic daily activities, measuring the reduction in adaptive abilities and functions |
| | caused by a decrease in the function of the body's systems and measuring a decrease in size and strength |
| | muscle) 1 week after the first examination. After the VR study is over, you will |
| | given a token of gratitude in the form of a patient care guide book. |
| 5. | Risks, side effects and management |
| | You may feel a little dizzy when using the VR system, but this is |
| | there are no risks and there are no significant side effects on the participation that will be undertaken by |
| | Sir/Madam/Brother. |
| 6. Ber | nefits |
| | The benefit that you will get is that you have the opportunity to use the system |
| | VR as a free medical rehabilitation therapy facility. |
| 7. | Compensation |
| | After the VR research is over, you will be given a token of thanks in the form of an agenda book. |
| | patient care guide. |
| 8. | Financing |
| | All components of the research are funded by the researcher through research grants and without any |
| | support from sponsors. |
| 9. | Confidentiality |
| | Sir/Madam/Brother, you will be explained about the research stages before the research begins. Identity |
| | Sir/Madam/Brother will be identified by initials and given a special code to maintain confidentiality. |
| | Sir/Madam/Brother. The data is stored on the research computer and can only be accessed by the research team. |
| | consisting of the main researcher, other researchers and research assistants. |

# 10. Obligations of research subjects





\_\_\_\_\_\_

As a research subject, you are obliged to follow the research rules or instructions. as written above. If there is anything that is not clear, you can ask further questions to research team. During the study, no other medication or herbal medicine was allowed other than those prescribed. by researchers.

#### 11. The right to refuse and withdraw

Your participation in this research is voluntary. You can refuse to participate or withdraw from this research at any time, either before the research ongoing or during the research. You do not have to participate in this research if you do not wish to do so. You must understand that even though Sir/Madam/Brother agrees to participate, Sir/Madam/Brother has the right to withdraw from this research. If you refuse to participate or withdraw from this research, This decision will not affect your relationship with me and will not affect you. impact on the service standards that apply in this hospital. I will give you the opportunity to you at the end of this explanation so that you can consider the decision that will be made. taken.

### 12. Post-trial access

Post-research access is a guarantee that after the research is over, both subjects/participants both the group given the experimental therapy and the control group will receive treatment best according to test results.

#### 13. Additional Information

Sir/Madam/Brother, you are given the opportunity to ask any questions that are unclear regarding this matter. this research. If at any time side effects occur or further explanation is needed, Mr./
Mothers/sisters can contact **Dr. Melinda Harini**, **Sp.KFR(K)** on HP no. +62 815-9635-765 and **Prasandhya Astagiri Yusuf**, **S.Si**, **MT**, **Ph.D** at the **Department of Medical Rehabilitation**, **General Hospital Dr. Cipto Mangunkusumo National Center**.





sculty of Medicine, University of Indonesis-Central Java Hospital

# **RESEARCH PARTICIPATION CONSENT SHEET**

All these explanations have been conveyed to me and all my questions have been answered by

[research teaml doctor]. I understand that if I need an explanation, I can ask

[name of researcher/ doctor]

Certificate of Consent

| | | W. Control of the Con |
|---|---|---|
| given the opportunity to ask | tions about this study. I have been a questions, and all my questions have agree to participate in this research | I confirm that the participant has been given the opportunity to ask questions about this study, and all questions have been answered truthfully. I confirm that consent has been given voluntarily. |
| Name of subject/guardian | | Dr. Melinda Harini, Sp.KFR-K |
| <br>Study participant signature | | Signature of researcher/approval requester |
| Dateyear | day/month/ | Date day/month/<br>year |
| Researcher Information: | | |
| Principal Investigator: | Dr. Melinda Harini, Sp.KFR(K) | |
| | Department of Medical Rehabilitation, Dr. Cipto M | langunkusumo National Central General Hospital |
| | +62 815-9635-765 | |
| esearchers: Prasandhya Astagiri Yusuf, S.Si, MT, Ph.D | | |
| | Medical Technology Cluster, Medical Technology Cluster, Indonesian Medical Education and Research Institution. | |
| | Jl. Salemba Raya No. 6 Jakarta, Indonesia. | |
| | +62 812-8459-4272 | |
| Researchers: | Dr. Amien Suharti, SpKFR | |
| | Department of Medical Rehabilitation, University | of Indonesia Hospital |
| | +62 815-9279-716 | |
| Researchers: | Dr. Budiati Laksmitasari, Sp.KFR | |
| | Department of Medical Rehabilitation, Dr. Cipto Mangunkusumo National Central General Hospital | |
| | +62 81511298554 | |
| Head of FKUI-RSCM Faculty of Medicine and Nursing: | Jalan Salemba 6, Central Jakarta, 10430 | |
| | Tel. No.: 021 3157008 | |
| | Email: ec_fkui@yahoo.com | |

Page 5 of 5 version 02 dated February 6, 2024 0995/rev00/KEP/2019